CLINICAL TRIAL: NCT06137742
Title: A PHASE 1 / 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF SINGLE ESCALATING DOSES OF PF-07868489 IN HEALTHY ADULT PARTICIPANTS AND, ADDITIONALLY, CLINICAL ACTIVITY OF REPEAT DOSES IN PARTICIPANTS WITH PULMONARY ARTERIAL HYPERTENSION
Brief Title: A Study to Learn About the Study Medicine Called PF-07868489 in Healthy Adult People and in People With Pulmonary Arterial Hypertension
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C5001001; 2024-514064-17-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary; high lung artery pressure
MeSH Terms: conditions — Pulmonary Arterial Hypertension

STUDY DESIGN:
Intervention Model Description: Part A is a sequential study. Part B is a parallel group study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Part A is an investigator- and participant-blind, sponsor-open, placebo-controlled, single ascending dose.
  Part B is a 24-week, randomized, double blind, placebo-controlled study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PF-07868489 (Experimental): single subcutaneous injection (Part A); 6 subcutaneous injections at regular intervals (Part B)
  Interventions: Drug: PF-07868489
- Placebo (Placebo Comparator): single subcutaneous injection (Part A); 6 subcutaneous injections at regular intervals (Part B)
  Interventions: Drug: Placebo for PF-07868489

INTERVENTIONS:
Drug: PF-07868489 — Experimental Treatment
  Arms: PF-07868489
Drug: Placebo for PF-07868489 — Placebo
  Arms: Placebo

SUMMARY:
The purpose of the study is to learn how the study medicine called PF-07868489 is tolerated and acts in healthy adult people and people with pulmonary arterial hypertension (PAH).

Part A:

An investigator- and participant-blind, sponsor-open, placebo-controlled, single ascending dose study to assess the safety, tolerability, and pharmacokinetics (PK) of PF-07868489 in healthy adult participants.

Part B:

A 24-week, randomized, double blind, placebo-controlled study to assess the safety, tolerability, PK, and pharmacodynamics (PD) of PF-07868489 in adult participants with PAH.

ELIGIBILITY:
Key Inclusion Criteria Part A:

* overtly healthy
* Body mass index (BMI) of 16 to 32 kg/m2; and a total body weight >50 kg.

Key Exclusion Criteria Part A:

* clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, infections or allergic disease.
* smoking more than 10 cigarettes (or equivalent) per day or smoking history ≥10 pack-years.

Key Inclusion Criteria Part B:

* diagnosis of pulmonary arterial hypertension (PAH)
* stable dose of standard of care PAH vasodilators
* BMI 16 to 40 kg/m2; and a total body weight >45 kg.
* 6MWD ≥ 150 and ≤ 450.
* Pre-randomization RHC documenting a minimum of PVR ≥ 400 dyn ∙sec/cm5.

Key Exclusion Criteria Part B:

* Any medical or psychiatric condition or laboratory abnormality.
* Stopped receiving pulmonary hypertension chronic general supportive therapy 90 days prior to Day 1.
* Pulmonary capillary wedge pressure > 15 mmHg on right heart catheterization (RHC) conducted during Screening.
* History of severe allergic or anaphylactic reaction or hypersensitivity to recombinant proteins or excipients in investigational product.
* Major surgery within 8 weeks prior to randomization.
* Participants who smoke more than 10 cigarettes (or equivalent) per day or has a smoking history ≥10 pack-years.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2023-11-17 (Actual); Primary Completion 2026-09-02 (Estimated); Study Completion 2026-09-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Day 113.
  Part A
Number of Participants With Change From Baseline in Laboratory Tests Results | Baseline up to Day 113
  Part A
Number of Participants With Vital Sign Abnormalities | Baseline up to Day 113
  Part A
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Parameters | Baseline up to Day 113
  Part A
Number of Participants with Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Day 253
  Part B
Number of Participants With Change From Baseline in Laboratory Tests Results | Baseline up to Day 253
  Part B
Number of Participants With Vital Sign Abnormalities | Baseline up to Day 253
  Part B
Number of Participants With Change From Baseline in Electrocardiogram (ECG) Parameters | Baseline up to Day 253
  Part B
Change From Baseline in Pulmonary Vascular Resistance (PVR) at Week24 | Baseline, Week 24
  repeated doses

SECONDARY OUTCOMES:
Area Under the Plasma Concentration-time Profile From Time Zero to the Time of Last Quantifiable Concentration (AUClast) | Pre dose, 8, 12, 24, 48,72,96,168,336 hours post dose
  single dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) | Pre dose, 8, 12, 24, 48,72,96,168,336 hours post dose
  single dose
Maximum Observed Plasma Concentration (Cmax) | Pre dose, 8, 12, 24, 48,72,96,168,336 hours post dose
  single dose
Time to Reach Maximum Observed Plasma Concentration (Tmax) | 4-7 days
  single dose
Incidence of Anti-Drug Antibody (ADA) | Baseline and up to week 16
  single dose
Plasma Decay Half-Life (t1/2) | Day 113
  single dose
Minimum Observed Plasma Trough Concentration (Cmin) | Day 253
  repeat doses
Plasma Decay Half-Life (t1/2) | Day 253
  repeat doses
Incidence of Anti-Drug Antibody (ADA) | Baseline and up to Day 253
  repeated doses
Change From Baseline in N-Terminal Prohormone Brain Natriuretic Peptide (NT-proBNP) Concentration at Week24 | Baseline, Week 24
  repeated doses
6MWD | Baseline, Week 24
  repeated doses

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (62):
- United States (22):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - UCI Health - Costa Mesa, Costa Mesa, California
  - UCI Health Center for Innovative Health Therapies (CIHT), Orange, California
  - University of California, Irvine Medical Center, Orange, California
  - UC Davis Health Medical Center, Sacramento, California
  - University of California Davis Health, Sacramento, California
  - UCSF Health St. Mary's Hospital, San Francisco, California
  - UCSF Helen Diller Medical Center at Parnassus Heights, San Francisco, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Norton Hospital, Louisville, Kentucky
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - Icahn school of medicine at Mount Sinai, New York, New York
  - Eastowne 100 Medical Office Building, Chapel Hill, North Carolina
  - Eastowne Medical Office Building - Clinical Research Unit, Chapel Hill, North Carolina
  - UNC Health - Eastowne Medical Office, Chapel Hill, North Carolina
  - UNC Hospitals, Chapel Hill, North Carolina
  - Investigational Drug Services Pharmacy, Morrisville, North Carolina
  - Rhode Island Hospital, Providence, Rhode Island
  - Center for Advanced Lung Care, Providence, Rhode Island
  - Medical University of South Carolina - Nexus, Charleston, South Carolina
  - Medical University of South Carolina - Radiology, Charleston, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
- Australia (2):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Wesley Research Institute, Auchenflower, Queensland
- Belgium (2):
  - Université Libre de Bruxelles - Hôpital Erasme, Brussels, Bruxelles-capitale, Région de
  - UZ Leuven, Leuven, Vlaams-brabant
- Canada (2):
  - London Health Sciences Centre - Verspeeten Family Cancer Centre, London, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
- China (4):
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality
- Czechia (2):
  - Vseobecna fakultni nemocnice v Praze, Prague
  - Institut Klinicke a Experimentalni Mediciny, Prague
- France (3):
  - CHRU de Brest, Brest, Finistère
  - Centre Hospitalier Universitaire de Saint Étienne - Hôpital Nord, Saint Priest En Jarez, Pays de la Loire Region
  - Chu Grenoble Alpes, La Tronche
- Germany (5):
  - Thoraxklinik-Heidelberg gGmbH, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Regensburg, Regensburg, Bavaria
  - UKGM Gießen/Marburg, Giessen, Hesse
  - Universitätsmedizin Greifswald, Greifswald, Mecklenburg-Vorpommern
  - Universitaetsklinikum Carl Gustav Carus, Technischen Universitaet Dresden, Dresden, Saxony
- University General Hospital "ATTIKON" - General Hospital of West Attica "H AGIA VARVARA", Chaïdári, Attikí, Greece
- Italy (3):
  - Fondazione IRCCS San Gerardo dei Tintori, Monza, Monza E Brianza
  - ISMETT Istituto Mediterraneo per i Trapianti e Terapie ad Alta Specializzazione, Palermo
  - Fondazione IRCCS Policlinico San Matteo, Pavia
- Japan (5):
  - Kobe University Hospital, Kobe, Hyōgo
  - St. Marianna University Hospital, Kawasaki, Kanagawa
  - Tohoku University Hospital, Sendai, Miyagi
  - Yokohama City University Hospital, Kanagawa
  - National Hospital Organization Okayama Medical Center, Okayama
- South Korea (4):
  - Gachon University Gil Medical Center, Namdong-gu, Incheon-gwangyeoksi [incheon]
  - Seoul National University Hospital, Seoul, Seoul-teukbyeolsi [seoul]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul-teukbyeolsi [seoul]
  - Samsung Medical Center, Seoul, Seoul-teukbyeolsi [seoul]
- Spain (3):
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario La Paz, Madrid, Madrid, Comunidad de
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (4):
  - Hammersmith Hospital, London, London, CITY of
  - Golden Jubilee National Hospital, Clydebank
  - Royal Free London NHS Foundation Trust, Royal Free Hospital, London
  - Royal Brompton Hospital, London

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C5001001